CLINICAL TRIAL: NCT00871403
Title: An Open-label, Multicentre, Randomised Phase II Study of Pazopanib in Combination With Pemetrexed in First-line Treatment of Subjects With Predominantly Non-squamous Cell Stage IIIBwet/IV Non-small Cell Lung Cancer
Brief Title: Study of Pazopanib and Pemetrexed in Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111128
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Results first posted 2012-02-16 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2012-03

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: GW786034; pazopanib; pemetrexed; cisplatin; non-small cell lung cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pazopanib; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Investigational treatment (pazopanib and pemetrexed)
  Interventions: Drug: pazopanib and pemetrexed
- Arm 2 (Active Comparator): Standard treatment (pemetrexed and cisplatin)
  Interventions: Drug: pemetrexed and cisplatin

INTERVENTIONS:
Drug: pazopanib and pemetrexed — oral pazopanib 600 mg once daily and pemetrexed intravenous (IV) 500mg/m^2 once every 3 weeks, then pazopanib 800 mg once daily
  Arms: Arm 1
Drug: pemetrexed and cisplatin — pemetrexed IV 500 mg/m^2 and cisplatin IV 75 mg/m^2 once every 3 weeks
  Arms: Arm 2

SUMMARY:
The main purpose of this study is to determine whether the combination of pazopanib and pemetrexed is safe and effective in the treatment of advanced non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* At least 18 years old
* Histologically- or cytologically-confirmed diagnosis of predominantly nonsquamous cell Stage IIIBwet (with confirmed malignant pleural effusion) or Stage IV NSCLC
* No prior systemic first-line therapy for advanced NSCLC
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of at least 12 weeks
* Able to swallow and retain oral medication
* Adequate organ system function (hematological, hepatic, and renal)
* Non-childbearing potential (i.e., physiologically incapable of becoming pregnant) OR childbearing potential, and agrees to use adequate contraception. A male with a female partner of childbearing potential is eligible if he uses a barrier method of contraception or abstinence during the study

Exclusion Criteria:

* Active malignancy or any malignancy in the 3 years prior to first dose of study drug other than NSCLC
* Central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for asymptomatic, previously treated CNS metastases
* Clinically significant gastrointestinal abnormalities
* Prolongation of corrected QT interval (QTc) > 480 msecs
* History of any one or more cardiovascular conditions within the past 6 months prior to randomization
* Poorly controlled hypertension
* History of cerebrovascular accident (including transient ischemic attacks), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months
* Major surgery or trauma within 28 days or any non-healing wound, fracture, or ulcer
* Evidence of active bleeding or bleeding diathesis
* Recent hemoptysis
* Endobronchial lesions and/or lesions infiltrating major pulmonary vessels
* Serious and/or unstable pre-existing medical (e.g., uncontrolled infection), psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures
* Use of any prohibited medication
* Use of an investigational agent within 28 days or 5 half-lives, whichever is longer, prior to the first dose of study drug
* Ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity except alopecia
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib, pemetrexed, and/or cisplatin
* Inability to interrupt aspirin or other non-steroidal anti-inflammatory drugs during the study
* Inability or unwillingness to take folic acid, vitamin B12 supplementation, or dexamethasone
* Clinically significant third-space fluid collections (e.g., ascites or pleural effusions) that cannot be controlled by drainage or other procedures prior to study start
* Recent or concurrent yellow fever vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2009-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Herlev, Denmark
- GSK Investigational Site, Sutton, Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, the study had 2 treatment arms: Arm 1, investigational (pazopanib+pemetrexed); and Arm 2, standard of care (cisplatin+pemetrexed). Protocol amendment 1 lowered the pazopanib starting dose (SD) for new Arm 1 participants from 800 to 600 milligrams. For clarity, safety/demography data for these different SDs are presented separately.
Groups:
- Pazopanib 600 mg Plus Pemetrexed 500 mg/m^2: Oral pazopanib 600 milligrams (mg) once daily plus intravenous pemetrexed 500 mg/meters squared (m^2) once every 3 weeks for 4 or 6 cycles during the Combination Treatment Phase.
- Pazopanib 800 mg Plus Pemetrexed 500 mg/m^2: Oral pazopanib 800 mg once daily plus intravenous (IV) pemetrexed 500 mg/ m^2 once every 3 weeks for 4 or 6 cycles during the Combination Treatment Phase. If participants experienced no disease progression, unacceptable toxicities, or death during the Combination Treatment Phase, they continued on pazopanib 800 mg monotherapy until disease progression, unacceptable toxicities, or death.
- Cisplatin 75 mg/m^2 Plus Pemetrexed 500 mg/m^2: IV cisplatin 75 mg/m^2 plus intravenous pemetrexed 500 mg/m^2 once daily every 3 weeks for 4 or 6 cycles during the Combination Treatment Phase. Until Protocol Amendment 2, upon disease progression participants had the opportunity to receive pazopanib 800 mg monotherapy if the investigator considered it an appropriate treatment option after considering alternative options for second-line treatment.
Period: Combination Treatment Phase
Arm/Group | Pazopanib 600 mg Plus Pemetrexed 500 mg/m^2 | Pazopanib 800 mg Plus Pemetrexed 500 mg/m^2 | Cisplatin 75 mg/m^2 Plus Pemetrexed 500 mg/m^2
Started | 9 | 62 | 35
Completed | 0 (No particiapants completed Combination Treatement.) | 13 (These participants completed combination treatment) | 23 (These participants completed combination treatment)
Not Completed | 9 | 49 | 12
Not completed — Randomized but Not Treated | 1 | 1 | 1
Not completed — Treatment Stopped; Protocol Amendment | 8 | 19 | 0
Not completed — Adverse Event | 0 | 17 | 2
Not completed — Disease Progression | 0 | 8 | 5
Not completed — Withdrawal by Subject | 0 | 3 | 1
Not completed — Physician Decision | 0 | 1 | 3
Period: Monotherapy Treatment Phase
Arm/Group | Pazopanib 600 mg Plus Pemetrexed 500 mg/m^2 | Pazopanib 800 mg Plus Pemetrexed 500 mg/m^2 | Cisplatin 75 mg/m^2 Plus Pemetrexed 500 mg/m^2
Started | 0 | 13 | 1
Completed | 0 | 0 | 0
Not Completed | 0 | 13 | 1
Not completed — Disease Progression | 0 | 9 | 1
Not completed — Adverse Event | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pazopanib 600 mg Plus Pemetrexed 500 mg/m^2 | Pazopanib 800 mg Plus Pemetrexed 500 mg/m^2 | Cisplatin 75 mg/m^2 Plus Pemetrexed 500 mg/m^2 | Total
Number analyzed (Participants) | 9 | 62 | 35 | 106
Age Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (14.32) | 60.8 (8.27) | 61.8 (9.35) | 61.1 (9.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 23 | 12 | 37
  Male | 7 | 39 | 23 | 69
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 0 | 1 | 0 | 1
  Asian - Central/South Asian Heritage | 1 | 0 | 0 | 1
  White - Arabic/North African Heritage | 0 | 2 | 2 | 4
  White - White/Caucasian/European Heritage | 8 | 59 | 33 | 100

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the interval between the date of randomization (date on which the investigator evaluated the participant and first determined he/she had disease progression) and the first occurrence of progressive disease (PD) or death from any cause. Per Response Evaluation Criteria in Solid Tumors (RECIST), version 1, PD is defined as a >=20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of >=1 new lesion).
Time Frame: Randomization until progression or death (up to 85 weeks)
Population: Intent-to-Treat (ITT) Population: all participants randomized to receive treatment and who were analyzed based on the assigned randomized treatment and not based on actual treatment received/not received. Participants who had neither progressed nor died were censored at the date of the last adequate tumor assessment at the time of the cut-off.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pazopanib 800 mg Plus Pemetrexed 500 mg/m^2 | Cisplatin 75 mg/m^2 Plus Pemetrexed 500 mg/m^2
Number analyzed (Participants) | 62 | 35
weeks | 25.0 [17.3 to 34.1] | 22.9 [18.4 to 27.7]
Statistical Analysis 1: Comparison: Pazopanib 800 mg Plus Pemetrexed 500 mg/m^2 vs Cisplatin 75 mg/m^2 Plus Pemetrexed 500 mg/m^2; Test type: Superiority or Other; p = 0.2647, Log Rank; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.43 to 1.28] — The hazard ratios is estimated using a Pike estimator. The estimated value is the hazard ratio comparing Pazopanib 800 mg plus pemetrexed 500 mg/m^2 to Cisplatin 75 mg/m^2 plus pemetrexed 500 mg/m^2

2. Secondary Outcome: Overall Survival (OS)
Description: OS was determined from the date of randomization to the date of death from any cause. Participants who had not died at the time of the cut-off for the final analysis were censored at the date the participants were last known to be alive. Because enrollment in the study was halted prematurely, the ability to achieve an estimate of OS was compromised. Consequently, OS was not estimated.
Time Frame: Randomization until death (up to 85 weeks)
Population: ITT Population
Arm/Group | Pazopanib 800 mg Plus Pemetrexed 500 mg/m^2 | Cisplatin 75 mg/m^2 Plus Pemetrexed 500 mg/m^2
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Best Overall Response, Assessed as the Number of Participants With the Indicated Tumor Response: Investigator Assessed Only
Description: Tumor response was assessed by the Investigator according to the RECIST, version 1.0. A participant was defined as a responder if he/she sustained a complete response (CR; the disappearance of all target lesions) or partial response (PR; >=30% decrease in the sum of the longest diameter of target lesions) for at least 4 weeks at any time during randomized treatment. Stable disease is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter since the treatment started.
Time Frame: Randomization until response or progressive disease (up to 85 weeks)
Population: ITT Population. A participant without a post-baseline assessment of response was considered to be a non-responder; i.e., all randomized participants are included in the denominator.
Measure: Number; unit: participants
Arm/Group | Pazopanib 800 mg Plus Pemetrexed 500 mg/m^2 | Cisplatin 75 mg/m^2 Plus Pemetrexed 500 mg/m^2
Number analyzed (Participants) | 62 | 35
participants
  Complete response | 0 | 0
  Partial response | 14 | 12
  Stable disease | 13 | 14
  Progressive disease | 6 | 5
  Unknown | 29 | 4

4. Secondary Outcome: Percentage of Participants With a Complete Response or a Partial Response
Description: The percentage of participants with a complete response or a partial response was evaluated.
Time Frame: Randomization until response or progressive disease (up to 85 weeks)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Pazopanib 800 mg Plus Pemetrexed 500 mg/m^2 | Cisplatin 75 mg/m^2 Plus Pemetrexed 500 mg/m^2
Number analyzed (Participants) | 62 | 35
percentage of participants | 14 | 12
Statistical Analysis 1: Comparison: Pazopanib 800 mg Plus Pemetrexed 500 mg/m^2 vs Cisplatin 75 mg/m^2 Plus Pemetrexed 500 mg/m^2; Test type: Superiority or Other; p = 0.2113, Binomial asymptotic; percent difference in response = -12.0, 95% CI 2-sided [-30.6 to 7.2] — The estimated value is the percent difference in the response rate comparing Pazopanib 800 mg plus pemetrexed 500 mg/m^2 to Cisplatin 75 mg/m^2 plus pemetrexed 500 mg/m^2

ADVERSE EVENTS:
Description: Serious adverse events (SAEs) and non-serious AEs are presented for the entire treatment period (Combination Treatment Phase followed by the Monotherapy Phase). SAEs and AEs were collected in the Safety Population, comprised all participants who had received at least one dose of both drugs within the assigned regimen.
Arm/Group | Pazopanib 600 mg Plus Pemetrexed 500 mg/m^2 | Pazopanib 800 mg Plus Pemetrexed 500 mg/m^2 | Cisplatin 75 mg/m^2 Plus Pemetrexed 500 mg/m^2
Serious Adverse Events (participants affected / at risk) | 3/8 | 34/61 | 12/34
Other Adverse Events (participants affected / at risk) | 7/8 | 59/61 | 32/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 600 mg Plus Pemetrexed 500 mg/m^2 (N=8) | Pazopanib 800 mg Plus Pemetrexed 500 mg/m^2 (N=61) | Cisplatin 75 mg/m^2 Plus Pemetrexed 500 mg/m^2 (N=34)
Neutropenia (Blood and lymphatic system disorders) | 0 | 5 | 1
Pneumonia (Infections and infestations) | 1 | 3 | 2
Alanine aminotransferase increased (Investigations) | 0 | 5 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 4 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Hepatic enzyme increased (Investigations) | 0 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 2 | 0
Bronchopneumonia (Investigations) | 0 | 2 | 0
Disease progression (General disorders) | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pyrexia (General disorders) | 1 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 2 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bilirubin conjugated increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Death (General disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Embolism venous (Vascular disorders) | 0 | 0 | 1
Empyema (Infections and infestations) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Necrotising fascitis (Infections and infestations) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pneumonitis chemical (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Tumour embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Vasculitis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 600 mg Plus Pemetrexed 500 mg/m^2 (N=8) | Pazopanib 800 mg Plus Pemetrexed 500 mg/m^2 (N=61) | Cisplatin 75 mg/m^2 Plus Pemetrexed 500 mg/m^2 (N=34)
Nausea (Gastrointestinal disorders) | 4 | 24 | 21
Diarrhoea (Gastrointestinal disorders) | 0 | 21 | 6
Vomiting (Gastrointestinal disorders) | 1 | 15 | 12
Abdominal pain (Gastrointestinal disorders) | 0 | 10 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 7 | 4
Constipation (Gastrointestinal disorders) | 2 | 7 | 11
Dyspepsia (Gastrointestinal disorders) | 1 | 5 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 4 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 3 | 4
Flatulence (Gastrointestinal disorders) | 0 | 1 | 2
Mucosal inflammation (General disorders) | 1 | 10 | 3
Asthenia (General disorders) | 3 | 7 | 10
Pyrexia (General disorders) | 0 | 7 | 7
Non-cardiac chest pain (General disorders) | 0 | 3 | 6
Oedema peripheral (General disorders) | 0 | 3 | 0
Pain (General disorders) | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 36 | 9
Leukopenia (Blood and lymphatic system disorders) | 1 | 13 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 8 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 6 | 7
Anaemia (Blood and lymphatic system disorders) | 2 | 5 | 10
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 13 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 8 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 11 | 5
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 5 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 4 | 3
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 4 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 3 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Alanine aminotransferase increased (Investigations) | 0 | 11 | 1
Weight decreased (Investigations) | 0 | 9 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 8 | 1
Blood bilirubin increased (Investigations) | 0 | 4 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 4 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 3 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 1 | 4
Transaminases increased (Investigations) | 1 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 2
Hypertension (Vascular disorders) | 2 | 18 | 4
Decreased appetite (Metabolism and nutrition disorders) | 3 | 13 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 9 | 4
Dysgeusia (Nervous system disorders) | 0 | 4 | 2
Headache (Nervous system disorders) | 0 | 4 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 4 | 1
Lacrimation increased (Eye disorders) | 0 | 6 | 4
Conjunctivitis (Eye disorders) | 0 | 2 | 2
Dry eye (Eye disorders) | 0 | 0 | 3
Sleep disorder (Psychiatric disorders) | 0 | 3 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 3
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 4
Urinary retention (Renal and urinary disorders) | 0 | 1 | 2
Fatigue (General disorders) | 0 | 24 | 10

LIMITATIONS AND CAVEATS:
Efficacy data were only summarized for the pazopanib (pazo.) 800 mg + pemetrexed (peme.) 500 mg/m^2 and the cisplatin 75 mg/m^2 + peme. 500 mg/m^2 arms due to the small sample size/short treatment duration in the pazo. 600 mg + peme. 500 mg/m^2 arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.